CLINICAL TRIAL: NCT05675007
Title: The Effects of a Colon-delivered Multivitamin Supplement on Brain Functioning and Its Relation With Immunometabolic and Intestinal Markers in Ageing: the COMBI Study
Brief Title: Effects of a Colon-delivered Multivitamin Supplement on Brain Functioning, Immunometabolic- and Intestinal Markers in Ageing
Acronym: COMBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Donders Centre for Cognitive Neuroimaging (Other)
Collaborators: Wageningen University and Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 3033003.02
Record Dates: First submitted 2022-10-24; First posted 2023-01-09 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-05

CONDITIONS: Cognitive Decline; Aging
Keywords: Intestinal health; Gut-brain axis
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: This randomized controlled trial has two parallel intervention arms. One group will daily consume a colon-delivered multivitamin supplement for 6 weeks. The other group will daily consume a placebo tablet for 6 weeks. Participants will we randomly assigned to one of the two groups.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Stratified 1 to 1 randomization will be automatically performed in Castor. Participant, Investigator and Outcome Assessor will not be aware of the treatment group. An independent researcher will have access to randomization details, and make sure the participant will receive the correct supplement type.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colon-delivered multivitamin supplement (Experimental): Within this arm, study subjects will consume a colon-delivered multivitamin supplement for 6 weeks. Subjects are instructed to consume the capsule daily during breakfast. The capsule must be taken orally with a glass of water.
  Interventions: Dietary Supplement: Colon-delivered multivitamin supplement
- Placebo (Placebo Comparator): Within this arm, study subjects will consume a placebo capsule for 6 weeks. Subjects are instructed to consume the capsule daily during breakfast. The capsule must be taken orally with a glass of water.
  Interventions: Dietary Supplement: Placebo capsule

INTERVENTIONS:
Dietary Supplement: Colon-delivered multivitamin supplement — Colon-delivered multivitamin supplement containing the following dose of the indicated vitamin: vitamin B2 (10 mg), vitamin B3 (4.0 mg), vitamin B6 (1.4 mg), vitamin B9 (400 μg), vitamin C (200 mg) and vitamin D3 (15ug). Vitamin capsules are filled with microcrystalline cellulose and magnesium stearate up to 200 mg. Control of release in the colon is achieved by the Eudragit S 100 coating layer technology that surrounds the vitamins contained in the core capsules.
  Arms: Colon-delivered multivitamin supplement
Dietary Supplement: Placebo capsule — Placebo capsule containing microcrystalline cellulose and magnesium stearate up to 200 mg. Placebo capsules are coated with the Eudragit S 100 coating layer.
  Arms: Placebo

SUMMARY:
COMBI is a multi-center, randomized controlled trial among 70 older adults at risk of cognitive decline. The main goal is to investigate the effect of a 6-week colon-delivered multivitamin supplementation on the gut-brain axis in older adults, by assessing changes in brain function as well as intestinal changes compared to placebo.

DETAILED DESCRIPTION:
Growing evidence indicates an important role for intestinal health in development of cognitive decline in ageing. Intestinal health, and especially the gut microbiome, is assumed to affect brain health and functioning via immunometabolic pathways captured in the gut-brain axis. However, it is unclear whether changes in intestinal health markers causally relate to cognitive decline in older adults and how. Nutritional interventions specifically targeting the gut were found beneficial for human cognition and brain function. An intervention based on colon-delivered vitamins (B2, B3, B6, B9, C, D3) is proposed to affect gut health using microbiome-dependent and independent pathways. In this study, it will be investigated whether this intervention affects neurocognition in ageing humans, to reveal causal gut-brain relationships in aging.Therefore, the primary goal of the COMBI study is to investigate the effect of a 6-week colon-delivered multivitamin supplementation on the gut-brain axis in older adults, by assessing changes in brain function as well as intestinal changes compared to placebo. Secondary, the effects of this 6-week colon-delivered multivitamin supplementation in older adults on the following parameters related to potential gut-brain pathways will also be investigated: (1) other relevant brain parameters, (2) other relevant intestinal parameters, (3) immunometabolic parameters related to gut-brain pathways, and (4) neuropsychological test battery scoring.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age between 60-75 years (at pre-screening)
* Fluency in Dutch (speaking, reading and writing)
* Score ≥2 points on the risk factor scale below based on self report:

  * BMI≥25 (1 point)
  * Physical inactivity (according to WHO guidelines) (1 point)
  * Hypertension (1 point)
  * Hypertension without medication (1 point)
  * Hypercholesterolemia (1 point)
  * Diabetes type II (1 point)
  * Mild cardiovascular disease (1 point)

Exclusion Criteria:

* Food allergies or other issues with the vitamins included in the supplement
* Concurrent participation in other intervention trials
* Clinical diagnosis of ≥1 of the following:

  * Stroke;
  * Neurological disease(s) (e.g. MCI, dementia, MS, Parkinson's, epilepsy);
  * Current malignant disease(s), with or without treatment;
  * Current psychiatric disorder(s) (e.g. depression, psychosis, bipolar episodes, eating disorder);
  * Symptomatic cardiovascular disease (e.g. stroke, angina pectoris, heart failure, myocardial infarction);
  * Revascularisation surgery in the last 12 months at pre-screening;
  * Gastrointestinal diseases (i.e., diarrhoea, Crohn's disease, ulcerative colitis, diverticulosis, stomach or duodenal ulcers) or having a history of gastrointestinal surgical events (e.g. stoma) that may influence the results of the study, as determined by the study team;
  * Visual impairment (e.g. blindness);
  * Hearing or communicative impairment.
* Use of antibiotics within the previous 3 months before the study start.
* Use of protonpump inhibitors within the study period (esomeprazole, lansoprazole, omeprazole, pantoprazole, rabeprazole)
* Not willing to refrain from taking other supplements (containing vitamin B2, B3, B6, B9, or C, prebiotic, or probiotic) that can interfere with the study outcomes, from at least 2 weeks before start of the intervention till the end of the intervention period.
* Answering "Yes" on ≥1 of the Donders Institute MRI safety screening protocol questions (see the 8 questions below):

  1. Are there metal objects located in your upper body? Exception: tooth-fillings and/or dental crowns.
  2. Are there metal splinters in your body, in particular within the eyes? For example: through labour work in the metal industry.
  3. Are there jewellery items or piercings that you are unable to take off?
  4. Have you had a brain surgery in the past?
  5. Are there active implants present? For example: pacemaker, neurostimulator, insulin pump, hearing aid (that is unable to be removed).
  6. Are there any medical plasters or patches that you can't or may not take off? For example: nicotine patch.
  7. Do you suffer from epilepsy?
  8. Do you suffer from claustrophobia?
* Cognitive impairment as determined by Telephone Interview for Cognitive Status (TICS-M1), performed during pre-screening before inclusion and defined as a score <23.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2024-05-02 (Actual)

PRIMARY OUTCOMES:
Change in brain activity during working memory | Change between Baseline (T0), Follow-up after 6 weeks (T1)
  Blood-oxygen level dependent activity in dlPFC and hippocampus during N-back fMRI task
Change in working memory performance | Change between Baseline (T0), Follow-up after 6 weeks (T1)
  Task accuracy during N-back fMRI task
Change in faecal short-chain fatty acids | Change between Baseline (T0), Follow-up after 6 weeks (T1)
  Total faecal short-chain fatty acid concentration measured by gas chromatograph mass spectrometry

SECONDARY OUTCOMES:
Change in brain myo-inositol levels (neuroimaging) | Change between Baseline (T0), Follow-up after 6 weeks (T1)
  Brain myo-inositol levels reflecting neuroinflammation in dlPFC and hippocampus, measured by magnetic resonance spectroscopy
Change in cerebral perfusion levels (neuroimaging) | Change between Baseline (T0), Follow-up after 6 weeks (T1)
  Cerebral perfusion levels measured by arterial spin labelling
Change in neuropsychological test-battery scoring | Change between Baseline (T0), Follow-up after 6 weeks (T1)
  Z-scoring on cognitive domains predominantly affected by cognitive ageing: executive function (incl. working memory), episodic memory and processing speed.
Change in microbiota profile (faecal) | Change between Baseline (T0), Follow-up after 6 weeks (T1)
  16S rRNA based profile of gut microbiota in faeces
Change in individual short-chain fatty acids profile (faecal) | Change between Baseline (T0), Follow-up after 6 weeks (T1)
  GCMS measurement to assess profile of individual SCFAs in faeces (acetic acid, formic acid, propionic acid, isobutyric acid, butyric acid, isovaleric acid, valeric acid, 4-methyl valeric acid, hexanoic acid, heptanoic acid)
Change in stool water content (faecal) | Change between Baseline (T0), Follow-up after 6 weeks (T1)
  Water content of stool, based on wet- and dry weight.
Change in stool pH (faecal) | Change between Baseline (T0), Follow-up after 6 weeks (T1)
  Faecal pH will be measured with a pH/redox meter in faeces
Change in stool redox potential (faecal) | Change between Baseline (T0), Follow-up after 6 weeks (T1)
  Redox potential will be measured with a pH/redox meter in faeces
Change in intestinal inflammation profile (faecal) | Change between Baseline (T0), Follow-up after 6 weeks (T1)
  Assay-based profile of intestinal inflammation measured in faeces
Change in C-reactive protein concentration (blood) | Change between Baseline (T0), Follow-up after 6 weeks (T1)
  hsCRP measured via finger prick analysis
Change in white blood cell count (blood) | Change between Baseline (T0), Follow-up after 6 weeks (T1)
  White blood cell count measured via finger prick analysis
Change in inflammation profile (blood) | Change between Baseline (T0), Follow-up after 6 weeks (T1)
  Assay-based profile of systemic inflammation measured in plasma
Change in intestinal integrity profile (blood) | Change between Baseline (T0), Follow-up after 6 weeks (T1)
  Assay-based profile of intestinal integrity measured in plasma
Change in anti-oxidant status profile (blood) | Change between Baseline (T0), Follow-up after 6 weeks (T1)
  Assay-based profile of anti-oxidant status and oxidative stress measured in plasma
Change in metabolic profile (blood) | Change between Baseline (T0), Follow-up after 6 weeks (T1)
  Assay-based profile of (energy) metabolism measured in plasma
Change in brain health profile (blood) | Change between Baseline (T0), Follow-up after 6 weeks (T1)
  Assay-based profile of brain health measured in plasma
Change in vitamin profile (blood) | Change between Baseline (T0), Follow-up after 6 weeks (T1)
  Assay-based profile of circulating vitamins from supplement measured in plasma

OTHER OUTCOMES:
Body mass index | Baseline (T0)
  Measured in kg/m^2
Waist circumference | Baseline (T0)
  Measured in cm
Hip circumference | Baseline (T0)
  Measured in cm
Blood pressure | Baseline (T0)
  Scores range from approximately (for diastolic) 60-120 and (for systolic) 100-180 mmHg, with higher scores indicating higher blood pressure.
Abdominal fat distribution | Baseline (T0)
  VAT(visceral adipose tissue)/SAT(subcutaneous adipose tissue) ratio based on abdominal MRI scan
Baseline Demographics and medical history (questionnaire) | Baseline (T0)
  Demographic information, medical history and medication use - qualitative assessment
4DKL (questionnaire) | Baseline (T0)
  (Psychosocial) complaints in daily life. Separate scores for distress (>10 moderate, >20 severe), depression (>2 moderate, >5 severe), anxiety (>3 moderate, >9 severe) and somatisation (>10 moderate, >20 severe)
EQ-5D-5L (questionnaire) | Baseline (T0)
  Quality of life. Scores range from 0-100, higher scores indicate better quality of life
Five Facet Mindfulness Questionnaire (questionnaire) | Baseline (T0)
  Self-assessment of mindfulness. Total scale ranges from 24 - 120, higher scores indicate more mindfulness
LIBRA (questionnaire) | Baseline (T0)
  Modifiable dementia risk using lifestyle for brain health. The score ranges from -5.9 (minimum score) to +12.7 (maximum score), with higher scores meaning a worse outcome (higher dementia risk)
Lubben Social Network Scale (questionnaire) | Baseline (T0)
  Social contact and perceived social support. The score ranges from 0 (minimum score) to 30 (maximum score), with higher scores meaning a better outcome (higher level of perceived social support)
SARC-F Sarcopenia questionnaire (questionnaire) | Baseline (T0)
  Sarcopenia. Scores range from 0 to 10 (i.e. 0-2 points for each component; 0 = best to 10 = worst).
Sedentary Behaviour Questionnaire (questionnaire) | Baseline (T0)
  Average hours and minutes of sedentary behavior a day, range from 0 to 24 hours. Higher scores (more hours) means a more sedentary behavior.
Change in Nutritional intake (questionnaire) | Change between Baseline (T0), Follow-up after 6 weeks (T1)
  Nutritional intake measured with a Food Frequency Questionnaire, assessing food intake of the past month, qualitative assessment
Change in Perceived Stress Scale (questionnaire) | Change between Baseline (T0), Follow-up after 6 weeks (T1)
  Stress perception. Total score, scale 0 - 40, higher scores indicate more perceived stress
Change in Pittsburgh Sleep Quality Index (PSQI) (questionnaire) | Change between Baseline (T0), Follow-up after 6 weeks (T1)
  Sleep quality. Total score ranging from 0 to 21 with the higher total score (referred to as global score) indicating worse sleep quality
Change in SQUASH (questionnaire) | Change between Baseline (T0), Follow-up after 6 weeks (T1)
  Physical activity. METs derived from the Ainsworth's compendium of physical activity will be used to classify physical activity intensity (<1.5METs- sedentary, 1.6-2.9 METs- light, 3.0-5.9METs- moderate, >6.0- vigorous physical activity).
Gastrointestinal symptoms questionnaire (questionnaire) | Baseline (T0)
  Gastrointestinal symptoms, qualitative assessment
Gastrointestinal symptoms questionnaire (questionnaire) | Follow-up after 6 weeks (T1)
  Gastrointestinal symptoms, qualitative assessment
Bristol stool chart (questionnaire) | Baseline (T0)
  Classification of faeces type, qualitative assessment
Bristol stool chart (questionnaire) | Follow-up after 6 weeks (T1)
  Classification of faeces type, qualitative assessment
Gut transit time | Baseline (T0)
  Gut transit time measured by blue muffin consumption and appearance in faeces
Gut transit time | Follow up after 6 weeks (T1)
  Gut transit time measured by blue muffin consumption and appearance in faeces
Change in Cognitive Failures Questionnaire (questionnaire) | Change between Baseline (T0), Follow-up after 6 weeks (T1)
  Subjective cognitive functioning. Score ranges from 0-100. A higher total score indicates more subjective cognitive failure.
Change in Cognitive Emotions Regulation Questionnaire (questionnaire) | Change between Baseline (T0), Follow-up after 6 weeks (T1)
  Cognitive coping strategies. Answers are scored on a 7-point Likert-type scale ranging from 1 (strongly disagree) to 7 (strongly agree). The scoring takes the average of all the scores in each subscale of cognitive reappraisal and expressive suppression
Change in Hospital Anxiety and Depression Scale (questionnaire) | Change between Baseline (T0), Follow-up after 6 weeks (T1)
  Anxiety and depression. Separate scores for anxiety (max 21) and depression (max 21). For each domain, a score >8 indicates psychiatric condition of anxiety or depression.
Change in Memory Self-Efficacy MIA (questionnaire) | Change between Baseline (T0), Follow-up after 6 weeks (T1)
  Self-evaluation and confidence of memory. Sum of Part 1 + Part 2A and B. Part 1: Strategy (scores 10 - 50, higher scores indicate more use of strategies), Part 2A: Subjective memory functioning, scores ranges from 23 - 115, with higher scores indicate better memory self-efficacy and 2B: Locus, scores ranges from 7 - 35, higher scores indicate better perceived personal control over remembering abilities.
Change in Starkstein Apathy Scale (questionnaire) | Change between Baseline (T0), Follow-up after 6 weeks (T1)
  Screen and measure apathetic symptoms. A higher total score (range 0-42) indicates more severe apathy, with a score greater than 14 or greater is indicative of clinical apathy
User experiences (questionnaire) | Follow up after 6 weeks (T1)
  User experiences of the supplement - qualitative assessment.
COVID status (questionnaire) | Baseline (T0)
  Vaccination status, COVID history - qualitative assessment.
COVID status (questionnaire) | Follow up after 6 weeks (T1)
  Vaccination status, COVID history - qualitative assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Esther Aarts, prof. dr., Principal Investigator — Radboud University, Donders Centre for Cognitive Neuroimaging
Locations (2):
- Netherlands (2):
  - Radboud University, Donders Centre for Cognitive Neuroimaging, Nijmegen, Gelderland
  - Wageningen University and Research, Division of Human Nutrition and Health, Wageningen, Gelderland